CLINICAL TRIAL: NCT03985722
Title: Phase I Clinical Trial of Olaratumab Plus Trabectedin in Advanced Soft-tissue Sarcoma Patients
Brief Title: Olaratumab Plus Trabectedin in Advanced Soft-tissue Sarcoma Patients Soft-tissue Sarcoma Patients
Acronym: OLATRASTS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS 58; 2017-004771-32 (EudraCT Number)
Record Dates: First submitted 2019-05-30; First posted 2019-06-14 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Sarcoma, Soft Tissue
Keywords: advanced soft-tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Trabectedin

STUDY DESIGN:
Intervention Model Description: The study is a phase I, non-randomised, one-armed, multicenter trial, open-label.
  The dose escalation rules include patients in blocks of 3 o 6 patient. Treatment is a combination of unlimited cycles of oralatumab and trabectedin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Unlimited cycles of Olaratumab and Trabectedin (Experimental): The study is a phase I, non-randomised, one-armed, multicenter trial, open-label,.
  The dose escalation rules include patients in blocks of 3 o 6 patient. Treatment is a combination of unlimited cycles of oralatumab and trabectedin.
  Interventions: Drug: Olaratumab and Trabectedin

INTERVENTIONS:
Drug: Olaratumab and Trabectedin — Dose escalation levels:
  LEVEL -1: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 0.9 mg/m2 D1 This is a security level in case level 0 causes DLT.
  LEVEL 0*: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 1.1 mg/m2 D1. * Dose starting level is 0.
  LEVEL 1: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 1.3 mg/m2 D1.
  LEVEL 2: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 1.5 mg/m2 D1.
  LEVEL 3**: Olaratumab 20 mg/kg C1D1 and C1D8 (induction) + Trabectedin 1.5 mg/m2 D1 and Olaratumab 15 mg/kg D1 and D8 (maintenance) + Trabectedin 1.5 mg/m2 D1
  **In LEVEL 3, Olaratumab dose of 20 mg/kg will be considered only for the first 2 doses (as induction doses, cycle 1 days 1 and 8). Then, the maintenance dose will be 15 mg/m2 for the rest of cycles.
  Other Names: Lartruvo and Yondelis

SUMMARY:
Phase I, multicentre clinical trial of olaratumab plus trabectedin in patients with advanced soft-tissue sarcoma.

Olaratumab plus trabectedin could be synergistic and with a manageable toxicity profile in advanced STS.

The study is a phase I, non-randomised, one-armed, multicenter trial, open-label.

The dose escalation rules include patients in blocks of 3 o 6 patient. Treatment is a combination of unlimited cycles of oralatumab and trabectedin.

Primary clinical study endpoint of phase I:

- Determine the maximum tolerated dose (MTD) or the recommended dose of olaratumab combined with trabectedin in advanced soft tissue sarcoma

Secondary clinical study endpoints:

* Objective Response Rate (ORR): ORR is defined as the number of subjects with a Best Overall Response (BOR) according to RECIST 1.1.
* Progression free survival (PFS): time to progression or death from treatment initiation.
* Overall survival (OS): Time from treatment initiation until death. Efficacy measured through tumor response according to Choi criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow-up until tumor progression.
* Correlation of clinical outcome with translational biomarkers.
* Quality of life (QoL) measured per QLQ-C30 questionnaire of EORTC

DETAILED DESCRIPTION:
PHASE I DESIGN

The number of evaluable patients to be included in this trial is 25. However 28 patients will be enrolled considering the possibility of 3 non-evaluable cases.

The dose escalation rules proceed as follows: escalating in cohorts of 3-6 patients per dose level. Three patients are treated at a given dose level. If at least 2 patients are observed to have dose-limiting toxicity (DLT), the prior dose level is defined as the maximum tolerable dosage (MTD) (unless only 3 patients have been treated at that level, in which case it is the tentative MTD). If 0 of the 3 patients are observed to have DLT, the dose level is escalated one step for the next cohort of 3 patients, and the process continues as above. If exactly 1 of the 3 patients treated show DLT, 3 additional patients are treated at the current dose level. If none of these additional 3 patients show DLT, the dose level is escalated for the next cohort of 3 patients, and the process continues as above; otherwise, the prior dose level is defined as the MTD.

Dose-limiting toxicity (DLT) is usually defined as cycle 1 grade 3 or above toxicity, excepting grade 3 neutropenia unaccompanied by either fever or infection. More specifically, for this clinical trial, DLT will be applied only to either of the following toxicities occurring during the first treatment cycle:

Hematological toxicity:

* Febrile neutropenia with documented Grade ≥3 infection or sepsis
* Grade 4 thrombocytopenia, or Grade 3 thrombocytopenia complicated by haemorrhage
* Grade 4 neutropenia lasting 7 days or longer

Non-hematological toxicities:

Grade 3-4 events, excluding:

* Nausea or vomiting without appropriate antiemetic treatment.
* Grade 3 transaminitis will not be considered Dose Limiting Toxicity unless this would entail a delay in the treatment administration. This Adverse Event (AE) is well known as secondary effect of trabectedin in the first two cycles and has no clinical impact.

Dose-escalation levels:

LEVEL -1: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 0.9 mg/m2 D1 This is a security level in case level 0 causes DLT.

LEVEL 0*: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 1.1 mg/m2 D1

LEVEL 1: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 1.3 mg/m2 D1

LEVEL 2: Olaratumab 15 mg/Kg D1 and D8 + Trabectedin 1.5 mg/m2 D1

LEVEL 3**: Olaratumab 20 mg/kg Cycle 1, Day 1 (C1D1) and Cycle 1, Day 8 (C1D8) (induction) + Trabectedin 1.5 mg/m2 D1 Olaratumab 15 mg/kg D1 and D8 (maintenance) + Trabectedin 1.5 mg/m2 D1

* Dose starting level is 0.

**In the LEVEL 3 Olaratumab dose of 20 mg/kg will be considered only for the first 2 doses (as induction doses, cycle 1 days 1 and 8)) and then, the maintenance dose will be 15 mg/m2 for the rest of cycles.

Each cycle encompasses 21 days. It is not allowed dose-escalation for one given patient.

For safety reasons the first patient will be followed for 1 week before any other patient can be enrolled, given than the combination of trabectedin and olaratumab hasn't been administered to any patient so far.

For the inclusion of the third patient in a given dose-level it is necessary to have all the safety information of the first cycle of the previous 2 patients included in the same dose-level. Before moving on to the next dose-level, at least three patients must have been followed during 3 weeks (1 cycle).

The proposed trabectedin dose-level escalation is supported by previous phase I trials focusing on trabectedin combination. In STS, the lowest level for trabectedin was 0.9 mg/m2 for combination with doxorubicin 60 mg/m2 and showed to be active61. With other antiangiogenic agents, combination produced prolonged cytopenias. Therefore, starting level 0 uses Trabectedin 1.1mg/m2.

* Tumor samples to be collected: The most recent archive tumor sample (1 block) must be donated for diagnosis confirmation and for biomarker analysis and another tumor sample after 2 cycles of olaratumab and trabectedin is also mandatory..

When feasible another tumor block should be collected after treatment.

* Translational study:

1. Evaluate the signalling pathways underlying the response to the combination of olaratumab and trabectedin in formalin-fixe, paraffin-embedded (FFPE) samples, from STS patients (HTG Molecular Oncology Biomarker Panel (OBP) Assay).
2. Correlate the potential predictive biomarkers (immunomodulatory signature) of the response to olaratumab and trabectedin, with clinic results, such as progression-free survival (PFS), overall survival (OS) and response assessment.
3. To correlate the activity of olaratumab plus trabectedin with gene expression profiling in 3-methylcholanthrene (3-MCA) fibrosarcoma immunocompetent mice models.

Samples:

1. FFPE samples (pre-treatment), before enrolment and after cycle 2. Both biopsies are mandatory. If the patient did not received any treatment in the last 6 months, previously to the enrolment, any biopsy taken within this period will be acceptable to the translational study.
2. When feasible, optionally for the patient, another tumor block should be collected after the end of treatment.
3. Peripheral blood samples taken at baseline, cycle 1 days 8, pre-cycle 2 day 2, pre-cycle 3 day 1 and after documented response of progression and after progression in 1 PAXgene tube and 2 BD Vacutainer® Cellular Preparation Tube (CPT)™.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent prior to performance of study specific procedures and must be willing to comply with treatment and follow-up.
2. Age: 18-80 years.
3. Histologic diagnosis of soft tissue sarcoma: liposarcoma (dedifferentiated and myxoid/round cell), leiomyosarcoma, undifferentiated pleomorphic sarcoma, synovial sarcoma confirmed, before enrolment confirmation, by central pathology review by a paraffin embedded tumor tissue.
4. Metastatic/advanced disease in progression in the last 6 months.
5. Patients had previously received at least anthracyclines if clinically indicated.

   Previous olaratumab administration is allowed.
6. Measurable disease according to RECIST 1.1 criteria.
7. ECOG Performance Status of 0-1.
8. Adequate hepatic, renal, cardiac, and hematologic function.
9. Laboratory tests as follows: Haemoglobin >9g/dl, Absolute neutrophil count ≥ 1,500/mm³, Platelet count ≥ 100,000/mm³, Total Bilirubin ≤ 1.5 mg/dL, PT≤ 1.5 ULN and INR ≤ 1.5, AST and ALT ≤ 2.5 times upper limit of normal, Creatinine

   ≤ 1.5 mg/dL Calcium ≤ 12 mg/dL and Blood glucose < 150 mg/dL, Urine protein assessment: <2+, and/or <3.5g protein/24h.
10. Left ventricular ejection fraction ≥ 50% by echocardiogram or MUGA scan.
11. Having a central venous portal is mandatory before treatment initiation.
12. Females of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment. Females of child-bearing potential and males and must agree to use highly effective contraceptive precautions during the trial and up to 6 months following the last dose of study drug. A highly effective method of birth control is defined as one that results in a low failure rate (that is, <1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner.

Exceptions: Females not of child-bearing potential due to surgical sterilization (at least 6 weeks following surgical bilateral oophorectomy with or without hysterectomy or tubal ligation) confirmed by medical history or menopause. A "postmenopausal woman" is a woman meeting either of the following criteria:

* spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (for example, oral contraceptives, hormones, gonadotropin releasing hormone, antiestrogens, selective estrogen receptor modulators (SERMs), or chemotherapy
* spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone (FSH) level >40 mIU/mL

Exclusion criteria:

1. More than 2 previous lines of chemotherapy for advanced disease. Previous trabectedin not allowed.
2. Hipersensitivity to olaratumab.
3. The following histologies are not included: Ewing Sarcoma, extraskeletal osteosarcoma, extraskeletal myxoid chondrosarcoma, Kaposi's sarcoma, rhabdomyosarcoma and gastrointestinal stromal tumor (GIST).
4. Uncontrolled intercurrent illness including (not limited to): symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] III/IV), unstable angina pectoris or coronary angioplasty, or stenting within 24 weeks prior to registration, unstable cardiac arrhythmia (ongoing cardiac dysrhythmias of NCI-CTCAE] version 5.0 Grade >= 2), known psychiatric illness that would limit study compliance, intra-cardiac defibrillators, known cardiac metastases, or abnormal cardiac valve morphology (>= Grade 3).
5. Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
6. Other disease or illness within the past 6 months, including any of the following:

   * Myocardial infarction
   * Coronary or peripheral artery bypass graft
   * Cerebrovascular accident or transient ischemic attack
   * Pulmonary embolism
7. The patient has electively planned or will require major surgery during the course of the study
8. Social situation that would preclude study compliance.
9. Prolonged QTc interval (i.e., QTc > 450 msec for males or QTc > 470 msec for females) on baseline ECG.
10. Hemorrhage ≥ Grade 3 in the past 4 weeks.
11. Females who are pregnant or breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or the recommended dose for phase II of Olaratumab plus Trabectedin. | Recruitment duration: 18 months
  There will be determined the security profile for each dose level.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | During recruitment and follow-up (30 months)
  Objective Response Rate (ORR): ORR is defined as the number of subjects with a Best Overall Response (BOR) according to RECIST 1.1.
Progression free survival (PFS) | During recruitment and follow-up (30 months)
  Time to progression or death from treatment initiation
Overall survival (OS) | During recruitment and follow-up (30 months)
  Time from treatment initiation until death
Efficacy as per Choi criteria | During recruitment and follow-up (30 months)
  Measured through tumor response according to Choi criteria. The evaluation criteria will be based on the identification of target lesions in baseline and their follow-up until tumor progression
Correlation of clinical outcome with translational biomarkers (See Translational Section) | During recruitment and follow-up (30 months)
  Correlation of clinical outcome with translational biomarkers (See Translational Section)
QoL | Recruitment duration: 18 months
  Measured per QLQ-C30 questionnaire of EORTC.

CONTACTS AND LOCATIONS:
Overall Officials: Javier MARTIN-BROTO, MD, Study Chair — University Hospital "Fundación Jiménez Díaz"
Locations (1):
- GEIS, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
We are open to Individual participant data (IPD). Whenever there is a researcher interested in OLATRASTS raw data results, please contact the Study Chief to comment on the objectives and agreement of this sharing.